CLINICAL TRIAL: NCT04108455
Title: Alternate Biomarkers for Better Management of Diabetes During Pregnancy and Prediction of Neonatal Complications in Pregnant Women With Diabetes
Brief Title: Biomarkers During Pregnancy
Status: Unknown | Type: Observational
Last Known Status: Active, not recruiting
Sponsor: Washington University School of Medicine (Other)
Collaborators: National Institutes of Health (NIH) (NIH)
Responsible Party: Sponsor
Other Study IDs: 201808125
Record Dates: First submitted 2019-09-25; First posted 2019-09-30 (Actual); Last update posted 2023-05-06 (Actual); Status verified 2023-05

CONDITIONS: Diabetes Mellitus in Pregnancy; Gestational Diabetes
MeSH Terms: conditions — Diabetes, Gestational

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Retrospective
Biospecimen Retention: Samples Without DNA — serum and plasma
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: Yes | Unapproved Device: Yes | US Export: No

GROUPS / COHORTS (2):
- With Diabetes: Pregnant women with diabetes - either diagnosed beforehand or diagnosed during gestation
  Interventions: Other: Specimens Collected
- Controls: Biobank samples will be obtained from similar age/BMI/ethnicity women who do not have evidence of diabetes.
  Interventions: Other: Specimens Collected

INTERVENTIONS:
Other: Specimens Collected — Serum will be collected from patients at multiple times during pregnancy for later analysis.

SUMMARY:
This study aims to obtain preliminary data for utility of alternate biomarkers for monitoring glucose control in diabetic women during pregnancy and/or predicting risk of adverse neonatal events in these women.

DETAILED DESCRIPTION:
This study aims to obtain preliminary data for utility of alternate biomarkers for monitoring glucose control in diabetic women during pregnancy and/or predicting risk of adverse neonatal events in these women. Our population is unique compared to published studies and contains significant numbers of African American women and overweight or obese women. Two of these markers have been examined in several other populations of pregnant women and have shown utility for both outcomes. However, the recommended levels of these markers need to be determined in specific populations as ethnicity and BMI affect the values. Values obtained in recruited women will be compared with biobank samples from women who have no evidence or history of diabetes. Additionally, two other potentially promising markers will be examined (beta-hydroxybutyrate and triglycerides). Both these analytes change during pregnancy and beta-hydroxybutyrate has shown correlation with large for gestational status or macrosomia in some studies. A combination of markers may be a better predictor of adverse neonatal outcomes than a single marker.

ELIGIBILITY:
Inclusion Criteria:

* All women included in the study will either have diabetes diagnosed before pregnancy or will have been diagnosed during pregnancy (GDM). We do not exclude minors, since in Missouri, they may consent to medical treatment without parental consent for medical issues relating to pregnancy,

Exclusion Criteria:

* No specific exclusion criteria will be used. BMI data will be collected and utilized to sort patients into various subgroups, but will not be used as exclusion criteria.

Ages: 14 Years to 48 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Child, Adult
Study Population: Our study population includes a large percentage of African Americans as well as a significant percentage of women with BMI ≥30. All women enrolled in the study will be pregnant and have been diagnosed with diabetes.
Sampling Method: Non-Probability Sample
Enrollment: 47 (Actual)
Dates: Start 2019-03-15 (Actual); Primary Completion 2021-11-01 (Actual); Study Completion 2023-11-30 (Estimated)

PRIMARY OUTCOMES:
Glucose Control | up to 60 weeks from enrollment
  various measures of glucose control will be reported and compared to other biomarkers measured by the study
Adverse Neonatal Events | up to 60 weeks from enrollment
  various adverse neonatal events will be reported and compared to other biomarkers measured by the study

SECONDARY OUTCOMES:
Glycated Albumin | up to 60 weeks from enrollment
  Levels of % glycated albumin will be measured in the various cohorts to see if correlations exist with glucose control and adverse neonatal events
Glycated Serum Protein (GSP) | up to 60 weeks from enrollment
  Levels of glycated serum protein will be measured in the various cohorts to see if correlations exist with glucose control and adverse neonatal events
Beta-hydroxybutyrate | up to 60 weeks from enrollment
  Levels of beta-hydroxybutyrate will be measured in the various cohorts to see if correlations exist with glucose control and adverse neonatal events
Triglycerides | up to 60 weeks from enrollment
  Levels of triglycerides will be measured in the various cohorts to see if correlations exist with glucose control and adverse neonatal events

CONTACTS AND LOCATIONS:
Overall Officials: Ebony Carter, MD, Study Chair — Washington University School of Medicine
Locations (1):
- Washington University in St Louis, St Louis, Missouri, United States

IPD SHARING:
Plan to Share IPD: No